CLINICAL TRIAL: NCT01644617
Title: A Phase IIb, Randomized, Placebo-Controlled, Dose-Finding Clinical Trial to Study the Safety and Efficacy of MK-8237 Using an Environmental Exposure Chamber in Subjects With House Dust Induced Allergic Rhinitis/Rhinoconjunctivitis
Brief Title: A Dose-Ranging Study of the Safety and Effectiveness of MK-8237 in the Treatment of House Dust Mite (HDM) Induced Allergic Rhinitis/Rhinoconjunctivitis in Adults (MK-8237-003/P07627)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P07627; 2012-001855-38 (EudraCT Number); 8237-003 (Other: Merck Registration Number)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Nonseasonal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo rapidly dissolving tablet administered sublingually once daily (q.d.), at approximately the same time each day, for 24 weeks
  Interventions: Drug: Placebo
- MK-8237 6 Developmental Units (DU) (Experimental): MK-8237 6 DU rapidly dissolving tablet administered sublingually q.d., at approximately the same time each day, for 24 weeks
  Interventions: Drug: MK-8237 6 DU
- MK-8237 12 DU (Experimental): MK-8237 12 DU rapidly dissolving tablet administered sublingually q.d., at approximately the same time each day, for 24 weeks
  Interventions: Drug: MK-8237 12 DU

INTERVENTIONS:
Drug: Placebo — Placebo rapidly dissolving tablets administered sublingually once daily
  Arms: Placebo
Drug: MK-8237 6 DU — MK-8237 6 DU rapidly dissolving tablets administered sublingually once daily
  Other Names: SCH 900237
  Arms: MK-8237 6 Developmental Units (DU)
Drug: MK-8237 12 DU — MK-8237 12 DU rapidly dissolving tablets administered sublingually once daily
  Other Names: SCH 900237
  Arms: MK-8237 12 DU

SUMMARY:
The purpose of this study is to evaluate the dose-related effectiveness, the safety and the tolerability of MK-8237, compared to placebo, in the treatment of house dust mite (HDM)-induced allergic rhinitis/rhinoconjunctivitis in adults. The primary hypothesis is that administration of MK-8237, compared to placebo, results in dose-related improvement in the average total nasal symptom score (TNSS) determined during environmental exposure chamber (EEC) challenge.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic rhinitis/rhinoconjunctivitis to house dust of 1 year duration or more (with or without asthma)
* If female of childbearing potential, has a negative urine pregnancy test at screening and agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control within the projected duration of the study.

Exclusion Criteria:

* Sensitized and regularly exposed to animal dander and molds, (e.g. present in the home, job, etc.)
* Sensitized and regularly exposed to seasonal allergens (i.e., birch or grass pollen)
* Immunosuppressive treatment within 3 months prior to screening (except steroids for allergic and asthma symptoms)
* History of chronic urticaria and/or angioedema within 2 years prior to screening
* Previous immunotherapy treatment with any HDM allergen for more than 1 month within 3 years prior to screening
* Ongoing treatment with any specific immunotherapy
* History of anaphylaxis with cardiorespiratory symptoms with prior immunotherapy, due to an unknown cause or to an inhalant allergen
* Unstable uncontrolled/partially controlled or severe asthma, or life-threatening asthma attack or an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids (but allowing short-acting beta agonists [SABA]) within 3 months prior to screening
* Asthma requiring medium- or high-dose inhaled corticosteroid (ICS) within 12 months prior to screening
* Chronic sinusitis within 2 years prior to screening
* Nasal condition that could confound the efficacy or safety assessments (e.g., nasal polyps)
* Pregnant, breastfeeding or planning to become pregnant during the study
* Participation in a different investigational study at any site during the same time frame of this study
* Direct association with the administration of the study or a family member of the study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Nolte H, Maloney J, Nelson HS, Bernstein DI, Lu S, Li Z, Kaur A, Zieglmayer P, Zieglmayer R, Lemell P, Horak F. Onset and dose-related efficacy of house dust mite sublingual immunotherapy tablets in an environmental exposure chamber. J Allergy Clin Immunol. 2015 Jun;135(6):1494-501.e6. doi: 10.1016/j.jaci.2014.12.1911. Epub 2015 Jan 27. PMID 25636947
- [Derived] Fortescue R, Kew KM, Leung MST. Sublingual immunotherapy for asthma. Cochrane Database Syst Rev. 2020 Sep 14;9(9):CD011293. doi: 10.1002/14651858.CD011293.pub3. PMID 32926419
- [Derived] Roth-Walter F, Schmutz R, Mothes-Luksch N, Lemell P, Zieglmayer P, Zieglmayer R, Jensen-Jarolim E. Clinical efficacy of sublingual immunotherapy is associated with restoration of steady-state serum lipocalin 2 after SLIT: a pilot study. World Allergy Organ J. 2018 Oct 1;11(1):21. doi: 10.1186/s40413-018-0201-8. eCollection 2018. PMID 30323863
- [Derived] Bernstein DI, Kleine-Tebbe J, Nelson HS, Bardelas JA Jr, Sussman GL, Lu S, Rehm D, Svanholm Fogh B, Nolte H. SQ house dust mite sublingual immunotherapy tablet subgroup efficacy and local application site reaction duration. Ann Allergy Asthma Immunol. 2018 Jul;121(1):105-110. doi: 10.1016/j.anai.2018.04.007. Epub 2018 Apr 12. PMID 29656145
- [Derived] Zieglmayer P, Nolte H, Nelson HS, Bernstein DI, Kaur A, Jacobi H, Lemell P, Schmutz R, Zieglmayer R, Horak F. Long-term effects of a house dust mite sublingual immunotherapy tablet in an environmental exposure chamber trial. Ann Allergy Asthma Immunol. 2016 Dec;117(6):690-696.e1. doi: 10.1016/j.anai.2016.10.015. PMID 27979028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants must have had a clinical history of allergic rhinitis/rhinoconjunctivitis (with or without asthma) to house dust of 1 year duration or more and determined to be sensitized to Dermatophagoides pteronyssinus and/or Dermatophagoides farina by skin prick test and immunoglobulin E levels. Other inclusion and exclusion criteria applied.
Groups:
- MK-8237 12 Development Units (DU): Participants received MK-8237 12 DU rapidly dissolving tablet administered sublingually once daily (q.d.), at approximately the same time each day, for 24 weeks.
- MK-8237 6 DU: Participants received MK-8237 6 DU rapidly dissolving tablet administered sublingually q.d., at approximately the same time each day, for 24 weeks.
- Placebo: Participants received placebo rapidly dissolving tablet administered sublingually q.d., at approximately the same time each day, for 24 weeks.
Period: Overall Study
Arm/Group | MK-8237 12 Development Units (DU) | MK-8237 6 DU | Placebo
Started | 42 | 41 | 41
Completed | 36 | 36 | 34
Not Completed | 6 | 5 | 7
Not completed — Withdrawal by Subject | 3 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 3 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8237 12 Development Units (DU) | MK-8237 6 DU | Placebo | Total
Number analyzed (Participants) | 42 | 41 | 41 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (9.2) | 26.7 (7.0) | 26.6 (6.1) | 26.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 30 | 17 | 66
  Male | 23 | 11 | 24 | 58

OUTCOME MEASURES:

1. Primary Outcome: Average Total Nasal Symptom Score (TNSS) During Environmental Exposure Chamber (EEC) Challenge Session at Week 24
Description: The average total TNSS included the evaluation of 4 nasal symptoms: itchy nose, blocked nose, runny nose, and sneezing. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 24. TNSS was the total of scores for the 4 nasal symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TNSS ranged from 0 to 12 points. The 24-week TNSS was analyzed using the analysis of covariance (ANCOVA) model with treatment and baseline TNSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TNSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 24
Population: Full Analysis Set including all randomized participants who received at least one dose of study treatment and had at least one post-randomization measurement for the analysis endpoint
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Groups:
- MK-8237 12 DU: Participants received MK-8237 12 DU rapidly dissolving tablet administered sublingually once daily (q.d.), at approximately the same time each day, for 24 weeks.
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 36 | 36 | 34
Score on a Scale | 3.83 [2.94 to 4.72] | 5.47 [4.55 to 6.39] | 7.45 [6.57 to 8.33]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Means (LSM) = -3.62, 95% CI 2-sided [-4.85 to -2.39] — Analysis by ANCOVA with treatment and baseline endpoint score as fixed effects and adjusted for different error variation for each treatment group
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Difference in LSM = -1.98, 95% CI 2-sided [-3.24 to -0.72] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Average TNSS During EEC Challenge Session at Week 16
Description: The average total TNSS included the evaluation of 4 nasal symptoms: itchy nose, blocked nose, runny nose, and sneezing. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 16. TNSS was the total of scores for the 4 nasal symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TNSS ranged from 0 to 12 points. The Week 16 TNSS was analyzed using the ANCOVA model with treatment and baseline TNSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TNSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 39 | 36 | 38
Score on a Scale | 4.82 [4.07 to 5.56] | 5.67 [4.83 to 6.50] | 6.90 [6.13 to 7.67]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LSM = -2.08, 95% CI 2-sided [-3.14 to -1.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.032, ANCOVA; Difference in LSM = -1.23, 95% CI [-2.36 to -0.11] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Average TNSS During EEC Challenge Session at Week 8
Description: The average total TNSS included the evaluation of 4 nasal symptoms: itchy nose, blocked nose, runny nose, and sneezing. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 8. TNSS was the total of scores for the 4 nasal symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TNSS ranged from 0 to 12 points. The Week 8 TNSS was analyzed using the ANCOVA model with treatment and baseline TNSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TNSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Score on a Scale | 5.34 [4.53 to 6.15] | 6.16 [5.55 to 6.78] | 6.71 [6.13 to 7.28]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA; Difference in LSM = -1.37, 95% CI 2-sided [-2.34 to -0.39] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.198, ANCOVA; Difference in LSM = -0.54, 95% CI 2-sided [-1.38 to 0.29] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Average Total Symptom Score (TSS [TNSS + TOSS]) During EEC Challenge Session at Week 24
Description: The average total TSS included the evaluation of the 4 nasal symptoms of the TNSS (itchy nose, blocked nose, runny nose, and sneezing) plus the 2 ocular symptoms of the TOSS (gritty/feeling/red/itchy eyes and watery eyes). The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 24. TSS was the total of scores for the 4 nasal symptoms and 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TSS ranged from 0 to 18 points. The Week 24 TSS was analyzed using the ANCOVA model with treatment and baseline TSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 36 | 36 | 34
Score on a Scale | 4.43 [3.20 to 5.66] | 6.62 [5.48 to 7.77] | 9.27 [7.98 to 10.57]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LSM = -4.84, 95% CI 2-sided [-6.59 to -3.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA; Difference in LSM = -2.65, 95% CI 2-sided [-4.35 to -0.95] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Average TSS (TNSS + TOSS) During EEC Challenge Session at Week 16
Description: The average total TSS included the evaluation of the 4 nasal symptoms of the TNSS (itchy nose, blocked nose, runny nose, and sneezing) plus the 2 ocular symptoms of the TOSS (gritty/feeling/red/itchy eyes and watery eyes). The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 16. TSS was the total of scores for the 4 nasal symptoms and 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TSS ranged from 0 to 18 points. The Week 16 TSS was analyzed using the ANCOVA model with treatment and baseline TSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 39 | 36 | 38
Score on a Scale | 5.95 [4.92 to 6.99] | 7.21 [6.05 to 8.37] | 8.58 [7.46 to 9.69]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LSM = -2.62, 95% CI 2-sided [-4.12 to -1.13] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.091, ANCOVA; Difference in LSM = -1.37, 95% CI 2-sided [-2.96 to 0.22] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Average TSS (TNSS + TOSS) During EEC Challenge Session at Week 8
Description: The average total TSS included the evaluation of the 4 nasal symptoms of the TNSS (itchy nose, blocked nose, runny nose, and sneezing) plus the 2 ocular symptoms of the TOSS (gritty/feeling/red/itchy eyes and watery eyes). The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 8. TSS was the total of scores for the 4 nasal symptoms and 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TSS ranged from 0 to 18 points. The Week 8 TSS was analyzed using the ANCOVA model with treatment and baseline TSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Score on a Scale | 6.51 [5.52 to 7.51] | 7.65 [6.81 to 8.48] | 8.48 [7.56 to 9.39]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA; Difference in LSM = -1.97, 95% CI 2-sided [-3.30 to -0.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.181, ANCOVA; Difference in LSM = -0.83, 95% CI 2-sided [-2.06 to 0.40] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Average Total Ocular Symptom Score (TOSS) During EEC Challenge Session at Week 24
Description: The average total TOSS included the evaluation of 2 ocular symptoms: gritty/feeling/red/itchy eyes and watery eyes. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 24. TOSS was the total of scores for the 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TOSS ranged from 0 to 6 points. The Week 24 TOSS was analyzed using the ANCOVA model with treatment and baseline TOSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TOSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 36 | 36 | 34
Score on a Scale | 0.61 [0.21 to 1.00] | 1.10 [0.68 to 1.53] | 1.87 [1.35 to 2.40]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LSM = -1.27, 95% CI 2-sided [-1.92 to -0.62] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.023, ANCOVA; Difference in LSM = -0.77, 95% CI 2-sided [-1.43 to -0.11] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Average TOSS During EEC Challenge Session at Week 16
Description: The average total TOSS included the evaluation of 2 ocular symptoms: gritty/feeling/red/itchy eyes and watery eyes. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 16. TOSS was the total of scores for the 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TOSS ranged from 0 to 6 points. The Week 16 TOSS was analyzed using the ANCOVA model with treatment and baseline TOSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TOSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 16
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 39 | 36 | 38
Score on a Scale | 1.14 [0.72 to 1.55] | 1.54 [1.05 to 2.03] | 1.67 [1.22 to 2.12]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p = 0.082, ANCOVA; Difference in LSM = -0.53, 95% CI 2-sided [-1.13 to 0.07] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.691, ANCOVA; Difference in LSM = -0.13, 95% CI 2-sided [-0.79 to 0.52] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Average TOSS During EEC Challenge Session at Week 8
Description: The average total TOSS included the evaluation of 2 ocular symptoms: gritty/feeling/red/itchy eyes and watery eyes. The endpoint was based on participant diary entries over the last 4 hours of the EEC challenge session at Week 8. TOSS was the total of scores for the 2 ocular symptoms, each scored on a 4-point rating scale (0=no symptoms; 1=mild symptoms; 2=moderate symptoms; 3=severe symptoms). The total TOSS ranged from 0 to 6 points. The Week 8 TOSS was analyzed using the ANCOVA model with treatment and baseline TOSS as covariates and expressed as a least squares mean with 95% confidence interval. A decrease in TOSS for participants receiving either dose of MK-8237 compared to placebo indicated an improvement in symptoms.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Score on a Scale | 1.18 [0.86 to 1.50] | 1.45 [1.08 to 1.83] | 1.79 [1.36 to 2.22]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p = 0.023, ANCOVA; Difference in LSM = -0.61, 95% CI 2-sided [-1.14 to -0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p = 0.235, ANCOVA; Difference in LSM = -0.34, 95% CI 2-sided [-0.90 to 0.22] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: HDM-specific Immunoglobulin E (IgE) Levels at Week 8
Description: Dermatophagoides pteronyssinus (D. pteronyssinus) and Dermatophagoides farinae (D. farinae) serum IgE levels were measured using the Immunocap® assay at Week 8. IgE levels were expressed in Log 10 scale kilo units/Liter (kU/L). Analysis was based on the analysis of variance parametric (ANOVA) model with treatment as the fixed effect and reported as mean IgE with a standard deviation.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log 10 kU/L
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Log 10 kU/L
  D. pteronyssinus | 1.77 (0.67) | 1.64 (0.53) | 1.25 (0.54)
  D. farinae | 1.80 (0.67) | 1.69 (0.53) | 1.31 (0.55)

11. Secondary Outcome: HDM-specific Immunoglobulin G4 (IgG4) Levels at Week 8
Description: D. pteronyssinus and D. farinae serum IgG4 levels were measured using the Immunocap® assay at Week 8. IgG4 levels were expressed in Log 10 scale milligrams/Liter (mg/L). Analysis was based on the ANOVA model with treatment as the fixed effect and reported as mean IgG4 with a standard deviation.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log 10 mg/L
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Log 10 mg/L
  D. pteronyssinus | -0.31 (0.40) | -0.33 (0.31) | -0.57 (0.11)
  D. farinae | -0.32 (0.47) | -0.31 (0.41) | -0.62 (0.22)

12. Secondary Outcome: Change From Baseline in HDM-specific IgE Levels at Week 8
Description: D. pteronyssinus and D. farinae serum IgE levels were measured using the Immunocap® assay at baseline and Week 8. IgE levels were expressed in Log 10 scale kU/L. Mean Week 8 IgE levels were compared to the mean IgE levels at baseline. Analysis was based on the ANOVA model with treatment as the fixed effect and reported as a least squares mean with 95% confidence interval.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Log 10 kU/L
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Log 10 kU/L
  D. pteronyssinus | 0.63 [0.51 to 0.75] | 0.50 [0.41 to 0.59] | 0.08 [0.03 to 0.12]
  D. farinae | 0.59 [0.48 to 0.70] | 0.46 [0.38 to 0.55] | 0.07 [0.03 to 0.11]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. pteronyssinus = 0.55, 95% CI 2-sided [0.43 to 0.68] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. pteronyssinus = 0.42, 95% CI 2-sided [0.33 to 0.52] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 3: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. farinae = 0.52, 95% CI 2-sided [0.41 to 0.64] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 4: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. farinae = 0.39, 95% CI 2-sided [0.30 to 0.48] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group

13. Secondary Outcome: Change From Baseline in HDM-specific IgG4 Levels at Week 8
Description: D. pteronyssinus and D. farinae serum IgG4 levels were measured using the Immunocap® assay at baseline and Week 8. IgG4 levels were expressed in Log 10 scale mg/L. Mean Week 8 IgG4 levels were compared to the mean IgG4 levels at baseline. Analysis was based on the ANOVA model with treatment as the fixed effect and reported as a least squares mean with 95% confidence interval.
Time Frame: Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Log 10 mg/L
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 40 | 39 | 39
Log 10 mg/L
  D. pteronyssinus | 0.23 [0.13 to 0.33] | 0.19 [0.12 to 0.25] | -0.00 [-0.01 to 0.01]
  D. farinae | 0.32 [0.22 to 0.41] | 0.24 [0.16 to 0.32] | -0.01 [-0.03 to 0.01]
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. pteronyssinus = 0.23, 95% CI 2-sided [0.13 to 0.33] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. pteronyssinus = 0.19, 95% CI 2-sided [0.12 to 0.25] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 3: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. farinae = 0.32, 95% CI 2-sided [0.23 to 0.42] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group
Statistical Analysis 4: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA; Difference in LSM: D. farinae = 0.25, 95% CI 2-sided [0.16 to 0.33] — Analysis by ANOVA with treatment as fixed effect and adjusted for different error variation for each treatment group

14. Secondary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. A serious adverse event (SAE) was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event.
Time Frame: From first dose to last dose of treatment plus 2 weeks of follow-up (Up to 26 weeks)
Population: All Participants as Treated including all randomized participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 42 | 41 | 41
Percentage of participants | 90.5 | 87.8 | 78.0
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; Difference in Percentage Versus Placebo = 12.4, 95% CI [-3.6 to 28.9] — Analysis based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; Difference in Percentage Versus Placebo = 9.8, 95% CI 2-sided [-7.0 to 26.6] — Analysis based on the Miettinen and Nurminen method

15. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: The percentage of participants who had study treatment stopped due to an AE. Discontinuations were reported for all randomized participants who received ≥1 dose of study treatment.
Time Frame: From first dose to last dose of treatment (Up to 24 weeks)
Population: All Participants as Treated including all randomized participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-8237 12 DU | MK-8237 6 DU | Placebo
Number analyzed (Participants) | 42 | 41 | 41
Percentage of Participants | 7.1 | 0.0 | 14.6
Statistical Analysis 1: Comparison: MK-8237 12 DU vs Placebo; Test type: Superiority or Other; Difference in Percentage Versus Placebo = -7.5, 95% CI 2-sided [-22.6 to 6.7] — Analysis based on the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: MK-8237 6 DU vs Placebo; Test type: Superiority or Other; Difference in Percentage Versus Placebo = -14.6, 95% CI 2-sided [-28.5 to -5.4] — Analysis based on the Miettinen and Nurminen method

ADVERSE EVENTS:
Time Frame: From first dose to last dose of treatment plus 2 weeks of follow-up (Up to 26 weeks)
Description: Adverse events collected for all randomized subjects who received at least one dose of study treatment
Arm/Group | MK-8237 12 Development Units (DU) | MK-8237 6 DU | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 1/41
Other Adverse Events (participants affected / at risk) | 36/42 | 35/41 | 24/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8237 12 Development Units (DU) (N=42) | MK-8237 6 DU (N=41) | Placebo (N=41)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8237 12 Development Units (DU) (N=42) | MK-8237 6 DU (N=41) | Placebo (N=41)
Ear pruritus (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 2 (2) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 8 (9) | 2 (2) | 1 (2)
Oedema mouth (Gastrointestinal disorders) | 10 (10) | 10 (10) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 6 (7) | 6 (6) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 12 (16) | 9 (11) | 8 (8)
Headache (Nervous system disorders) | 7 (9) | 6 (9) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 8 (13) | 13 (22)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 6 (7)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 14 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results without the prior written consent of the sponsor. The Sponsor has the opportunity to review all proposed abstracts, manuscripts, presentations, or data analyses regarding this trial 45 days prior to submission for publication/presentation. The sponsor has the right to review and comment with regard to proprietary information, accuracy, and compliance with FDA regulations.